CLINICAL TRIAL: NCT02861352
Title: Testing Novel Biomarkers of Zinc Status for Use in Human Zinc Supplementation Trials
Brief Title: An Evaluation of Zinc Status Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHO14
Record Dates: First submitted 2016-08-04; First posted 2016-08-10 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Inflammation; Oxidative Stress
Keywords: Zinc; DNA Integrity; Gene Expression; diet zinc; nutrition requirements
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diet zinc (Experimental): 3 dietary zinc levels: 6 mg/d, 10 mg/d and 25 mg supplemental zinc/d
  Interventions: Other: Diet zinc

INTERVENTIONS:
Other: Diet zinc — 4 mg zinc, as zinc sulfate, was added to a controlled diet; 25 mg supplemental zinc was given during the final recovery period when an ad lib diet was consumed

SUMMARY:
The purpose of this study is to determine the effect of a moderate decrease in dietary zinc on DNA strand breaks and other cellular zinc biomarkers.

DETAILED DESCRIPTION:
Assessing the zinc status of humans has proven to be difficult because of the unique physiological features of zinc homeostasis. Animal and human studies show that a small, vulnerable pool of cellular zinc is sensitive to changes in dietary zinc. The protein, Metallothionein (MT), is made within cells to stabilize this transient zinc pool and to provide a means to 'park' a small zinc reserve. The overall goal is to develop a new method for measuring MT in cells and to assess other cellular responses to changes in small changes in dietary zinc. Culture models of zinc deficiency and excess have been developed and used to test the response of cellular MT levels and mineralization to changes in zinc availability. In Phase II, the changes in the expression of leukocytic zinc transporters and the cellular in vitro uptake of isotopic zinc will be measured. Healthy men will be recruited to participate in a 6-week feeding trial to be followed by a 3-week recovery period. The results of this study will determine if potential new cellular zinc biomarkers respond to changes in zinc status when the men are fed an additional 4 mg zinc/d incorporated into a rice-based meal. These findings will provide essential, new information for designing an efficacy trial of biofortified rice and the zinc status of infants and young children.

ELIGIBILITY:
Inclusion Criteria:

* willing to limit food and beverage intake to that provided by the study
* willing to discontinue consumption of alcoholic beverages during the study
* has an operative understanding of English
* no plans to move from the area during the study period

Exclusion Criteria:

* chronic or acute metabolic disease (i.e., diabetes or asthma)
* taking medications for a metabolic disorder
* evidence of alcohol abuse or use of illicit drugs

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in the percent of leukocytic DNA strand breaks | Change in DNA strand breaks measured at baseline, 2, 4, and 3 week intervals with changes in diet zinc
  Baseline measurements were made upon entry into the study. Subsequent measurements were made after 2 weeks on a low zinc diet (6 mg/d), 4 weeks on a moderate zinc intake (10 mg/d) and after 3 weeks of consuming a 25 mg zinc supplement.

SECONDARY OUTCOMES:
Cellular zinc biomarkers | At baseline and at 3 time points during the 9 week study: after 2, 6, and 9 weeks.
  Specific measurements included the gene expression of zinc transporters, the in vitro uptake of leukocytic radioactive Zn, and a comprehensive serum metabolomic and proteomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Janet C King, Ph.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital Oakland Research Institute, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zyba SJ, Shenvi SV, Killilea DW, Holland TC, Kim E, Moy A, Sutherland B, Gildengorin V, Shigenaga MK, King JC. A moderate increase in dietary zinc reduces DNA strand breaks in leukocytes and alters plasma proteins without changing plasma zinc concentrations. Am J Clin Nutr. 2017 Feb;105(2):343-351. doi: 10.3945/ajcn.116.135327. Epub 2016 Dec 21. PMID 28003206